CLINICAL TRIAL: NCT05267197
Title: 3D Telemedicine: Communication During Covid 19. A Clinician Feedback Study
Brief Title: 3D Telemedicine: A Clinician Feedback Study
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Strathclyde (Other); Microsoft Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GN20HS181
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-02

CONDITIONS: Telemedicine; 3 Dimensional; Reconstructive Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D Telemedicine: Clinical consultation conducted with 3D Telemedicine
  Interventions: Other: 3D Telemedicine
- 2D Telemedicine: Clinical consultation conducted with 2D Telemedicine
  Interventions: Other: 2D Telemedicine

INTERVENTIONS:
Other: 3D Telemedicine — 3D Telemedicine system
  Groups: 3D Telemedicine
Other: 2D Telemedicine — 2D Telemedicine system
  Groups: 2D Telemedicine

SUMMARY:
The use of Telemedicine has increased significantly due to constraints imposed by the Covid pandemic. 3D telemedicine uses multiple cameras in the clinic room which can reconstruct an image in 3 dimensions in real-time, which may be beneficial in more visual focused specialties such as Plastic Surgery. There are no clinical data regarding the use of 3D telemedicine, with previous studies laboratory based without clinicians or patients. This study aims to provide clinician data comparing 3D and 2D Telemedicine, and feedback to allow incremental improvement of the system prior to clinical trials involving patients.

DETAILED DESCRIPTION:
Aims The aim of this study is to assess 3D telemedicine and 2D telemedicine from the clinician's perspective, to optimise the system prior to clinical trials with patients. This will provide baseline validated outcome data on areas such as usability, presence (the realism or immersion of a system), mental effort and task load. "Keep, Lose and Change" prompts will be used to aid improvements in the 3D Telemedicine system prior to clinical trials.

Participants This will be a clinician feedback based study on 2D telemedicine and 3D telemedicine. Clinicians will include nurses, doctors and physiotherapists from Canniesburn Plastic Surgery Unit, Glasgow, UK.

Consent Clinicians will consent in writing to participate

Method Clinicians will use both 3D and 2D Telemedicine systems to examine a member of the research team who will act as a "patient". There will be a single clinician (consultant, nurse specialist or physiotherapist) examining the patient during the clinic.They will use each system for 10 minutes each. No randomisation will take place. This will be followed by a questionnaire which will be filled in once per patient by the clinician in the clinic.

Outcome measures No primary or secondary measures are specified as this is an observational feedback study, not an interventional clinical trial.

Satisfaction - Visual Analogue Scale 0-100 Mental Effort Rating Scale - single instrument Likert scale (Paas 1996) System Usability Scale - 10 item industry standard technology scale Presence Questionnaire - 29 item scale - assessment of presence in the system/virtual environment (PQ, Witmer 2005).

Semi Structured exit interview - will discuss with participant their views on the telemedicine system, using "Keep, Lose and Change" prompts to aid system improvements.

ELIGIBILITY:
Inclusion Criteria:

* clinicians in Canniesburn Plastic Surgery Unit
* doctors
* nurses
* physiotherapists

Exclusion Criteria:

* visual problems whereby participant is legally blind
* cannot consent

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a mix of clinicians from Canniesburn Plastic Surgery Unit including:
  * doctors
  * nurses
  * physiotherapists These clinicians will be at varying levels of seniority, age and will be gender balanced, to provide generalisability of the results
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Clinical Satisfaction | 1 day (Single time point post study)
  Satisfaction measured on a Visual Analogue Scale between 0-100. Higher is better (Voutilainen et al. 2016).

SECONDARY OUTCOMES:
System Usability Scale | 1 day (Single time point post study)
  10 item industry standard technology scale, scores converted to a 0-100 scale. Higher is better
Presence Questionnaire | 1 day (Single time point post study)
  29 item scale - assessment of presence in the system/virtual environment. Score 0-203, Higher is better (PQ, Witmer 2005).
Mental Effort Rating Scale | 1 day (Single time point post study)
  Single instrument Likert scale rated 1-9. Lower is better (Paas 1996)

CONTACTS AND LOCATIONS:
Locations (1):
- Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD available on reasonable written request

REFERENCES:
- [Derived] Lo S, Fowers S, Darko K, Spina T, Graham C, Britto A, Rose A, Tittsworth D, McIntyre A, O'Dowd C, Maguire R, Chang W, Young D, Hoak A, Young R, Dunlop M, Ankrah L, Messow M, Ampomah O, Cutler B; 3DTM (3D Telemedicine) Collaborative research group; Armstrong R, Lalwani R, Davison R, Bagnall S, Hudson W, Shepperd M, Johnson J. Participatory development of a 3D telemedicine system during COVID: The future of remote consultations. J Plast Reconstr Aesthet Surg. 2023 Dec;87:479-490. doi: 10.1016/j.bjps.2022.10.012. Epub 2022 Oct 13. PMID 36890078